CLINICAL TRIAL: NCT02395796
Title: Efficacy of the Presence of a Pulsatile Pressure Waveform to Confirm Correct Placement of the Epidural Needle and Catheter in Laboring Pregnant Patients: a Feasibility Study
Brief Title: Pulsatile Pressure Waveform to Confirm Correct Placement of the Epidural in Laboring Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Negative results were obtained in all subjects that were analyzed (n=10)
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ilana Sebbag, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 106323
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Analgesia, Epidural
Keywords: epidural; labor analgesia; pressure monitoring
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epidural Pressure Waveform (Experimental): Study Population:
  * Term pregnancy
  * in labour
  * 18 years of age or older.
  Interventions: Procedure: Epidural Pressure Waveform

INTERVENTIONS:
Procedure: Epidural Pressure Waveform — When loss of resistance occurs, a high-pressure tubing extension will be connected to the needle and the pressure will be transduced and the waveform, recorded. An epidural catheter will then be passed through the needle and connected to a high-pressure tubing extension and the pressure will be transduced and recorded. A test dose of 3 mL of 2% lidocaine with epinephrine 1:200.000 will then be given to exclude potential spinal or intravascular injection. After 3 minutes, a loading dose of 10 mL of 0,125% bupivacaine will be given for labor analgesia and the presence or absence of a bilateral sensorial block at T10 or higher at 30 min will be assessed.

SUMMARY:
Epidural analgesia is highly effective for labor pain relief and is widely chosen by pregnant patients. However, placement of the epidural needle can be challenging in pregnant patients due to lax tissue ligaments and edema so that the traditional loss of resistance method (LOR) used to find the space may be subtle leading to retries which may delay onset of analgesia as well as increase the risk of complications. The ability to transduce a pulsatile pressure waveform from epidural needles placed in non-laboring patients correlates highly with successful placement of the epidural needle. We wish to evaluate the efficacy of obtaining a pulsatile pressure waveform with correct epidural needle placement in laboring women.

DETAILED DESCRIPTION:
Patients requesting epidural labor analgesia will be eligible for recruitment. After written informed consent is obtained, placement of monitors and aseptic technique, the 17G epidural needle will be placed using the loss of resistance (LOR) technique to air or saline at the lumbar level chosen by the anesthesiologist. When LOR occurs, the needle will then be filled with 2 mL NaCl 0.9% from that syringe and the pressure monitoring accessory will be connected to the needle. The second investigator will then connect the high pressure tubing to the acessory without touching it, and the pressure will be zeroed at level of the needle insertion. Pressure will then be transduced and the waveform, recorded. An epidural catheter (SIMS Portex) will then be passed through the needle and advanced 5 cm beyond the tip of the epidural needle. After securing the epidural catheter in place, the patient will be placed on the lateral position. The catheter will then be filled NaCl 0.9% from a syringe and a high-pressure tubing extension leveled at the spine level will be connected to the catheter and the pressure will be transduced and recorded. Data recorded will include 2 parameters: 1) The presence or absence of a pulsatile waveform, and 2) The actual pressure read at the epidural space, in mmHg. Those readings will be obtained in 2 distinct moments: at a " rest" state, meaning during an interval between contractions, and at an "active" state, during the first contraction after the epidural catheter is placed. A test dose of 3 mL of 2% lidocaine with epinephrine1:200.000 will then be given to exclude potential spinal or intravascular injection. After 3 minutes, a loading dose of 10mL of 0,125% bupivacaine will be given for labor analgesia and the presence or absence of a bilateral sensorial block at T10 or higher at 30 min will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients
* ASA I-III
* Term Pregnancy (>37 weeks)
* 18 years or older
* Early Labour (<6 cm of cervical dilation)
* BMI<40

Exclusion Criteria:

* Any contraindication to epidural analgesia placement (coagulopathy, sepsis, infection at site, increased ICP, hypovolemia, unstable ischemic heart disease, unstable neurologic disease, severe aortic stenosis, prior spinal surgery, LA allergy)
* Serious concern for maternal or fetal wellfare.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Epidural Needle Insertion Success | 30 min after loading dose
  Presence of a pulsatile pressure waveform at the epidural needle as a good predictor of a successful epidural block 30 min after local anesthetic injection

SECONDARY OUTCOMES:
Epidural Pressure in mmHg | 5 min after epidural needle insertion
  Epidural pressures during uterine contractions and in-between contractions in mmHg
Epidural Waveform at the Catheter | Immediately after epidural catheter insertion
  Presence or absence of an epidural waveform measured through the epidural catheter right after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, MD, FRCPC, Principal Investigator — University of Western Ontario, Schulich School of Medicine, Department of Anesthesia
Locations (1):
- Victoria Hospital- LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narang VP, Linter SP. Failure of extradural blockade in obstetrics. A new hypothesis. Br J Anaesth. 1988 Mar;60(4):402-4. doi: 10.1093/bja/60.4.402. PMID 3355735
- [Background] Ghia Jn, Arora Sk, Castillo M, Mukherji Sk. Confirmation of location of epidural catheters by epidural pressure waveform and computed tomography cathetergram. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):337-41. doi: 10.1053/rapm.2001.23932. PMID 11464353
- [Background] Lennox PH, Umedaly HS, Grant RP, White SA, Fitzmaurice BG, Evans KG. A pulsatile pressure waveform is a sensitive marker for confirming the location of the thoracic epidural space. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):659-63. doi: 10.1053/j.jvca.2006.02.022. Epub 2006 May 30. PMID 17023284
- [Background] Gong Y, Shi H, Wu J, Labu D, Sun J, Zhong H, Li L, Xin X, Wang L, Wu L, Ma D. Pressure waveform-guided epidural catheter placement in comparison to the loss-of-resistance conventional method. J Clin Anesth. 2014 Aug;26(5):395-401. doi: 10.1016/j.jclinane.2014.01.015. Epub 2014 Aug 27. PMID 25172504
- [Background] de Medicis E, Tetrault JP, Martin R, Robichaud R, Laroche L. A prospective comparative study of two indirect methods for confirming the localization of an epidural catheter for postoperative analgesia. Anesth Analg. 2005 Dec;101(6):1830-1833. doi: 10.1213/01.ANE.0000184130.73634.BE. PMID 16301268
- [Background] Messih MN. Epidural space pressures during pregnancy. Anaesthesia. 1981 Aug;36(8):775-82. doi: 10.1111/j.1365-2044.1981.tb08815.x. PMID 7294338
- [Background] Sivakumaran C, Ramanathan S, Chalon J, Turndorf H. Uterine contractions and the spread of local anesthetics in the epidural space. Anesth Analg. 1982 Feb;61(2):127-9. PMID 7198872